CLINICAL TRIAL: NCT05492032
Title: Cumulative and Booster Effects of Multisession Prefrontal Transcranial Direct-Current Stimulation (tDCS) on Cognitive and Social Impairments in Adolescents With Autism Spectrum Disorder
Brief Title: Cumulative and Booster Effects of Multisession Prefrontal Transcranial Direct Current Stimulation in Adolescents With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20220216004-01
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Transcranial Direct Current Stimulation; Autistic Spectrum Disorder; Electroencephalography; Booster Effects
Keywords: Autism; ASD; tDCS; Treatment outcome; EEG; E/I ratio; Booster effects; Cognitive function
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: This is a one-year parallel design (triple-arm), double-blind RCT. Participants will be randomly assigned to receive either (1) active daily tDCS with computerized executive function training in weeks 0-2, followed by active bimonthly booster tDCS sessions in weeks 3-14, and active monthly booster tDCS sessions in weeks 15-52; (2) active daily tDCS with computerized executive function training in weeks 0-2, followed by sham bimonthly booster tDCS sessions in weeks 3-14, and sham monthly booster tDCS sessions in weeks 15-52, or sham daily tDCS with computerized executive function training in weeks 0-2, followed by sham bimonthly booster tDCS sessions in weeks 3-14, and sham monthly booster tDCS sessions in weeks 15-52.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active cathodal (inhibitory) tDCS vs. Sham-tDCS condition (Experimental): Experimental group: active multisession tDCS + active booster tDCS vs Active control group: sham multisession tDCS + sham booster tDCS
  To test whether active cathodal [inhibitory] tDCS over the left dlPRC will facilitate learning through stimulation and thus improve cognitive function in patients with ASD, the primary outcomes (SRS-2 scores) of the two groups at the start (T0), 1-month (T1), 3-month (T2), 6-month (T3), and at the end of study i.e. 12-months (T4) will be compared.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS; Behavioral: Cognitive training
- Active booster tDCS treatment vs. Sham booster tDCS treatment (Experimental): Experimental group: active multisession tDCS + active booster tDCS vs Active control group: active multisession tDCS + sham booster tDCS
  To test whether booster treatment cycles of tDCS will prolong the cognitive benefits in individuals with ASD), the primary outcome, the total SRS-2 score, and the secondary outcomes, the E/I ratio and the cognitive composite score at the start (T0), 1-month (T1), 3-month (T2), 6-month (T3), and at the end of study i.e. 12-months (T4), will be compared.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS; Behavioral: Cognitive training
- Change in EEG E/I ratios in the active tDCS vs. sham tDCS groups (Experimental): Experimental group: active multisession tDCS + active booster tDCS vs Active control group: sham multisession tDCS + sham booster tDCS
  To test whether enhanced neuronal network organization, as indicated by EEG E/I ratios, in patients with ASD will mediate the beneficial effects of tDCS in terms of improvements in cognitive function, measurements taken at baseline, 1-day and 1-month after tDCS treatment will be compared. The change in EEG E/I ratios in patients in the active tDCS and sham tDCS groups will be compared using E/I ratios averaged from channels Fp1, F3, and F7 to increase the signal-to-noise ratio of the EEG data and to represent the left frontal E/I ratio.
  Interventions: Device: Active-tDCS; Device: Sham-tDCS; Behavioral: Cognitive training

INTERVENTIONS:
Device: Active-tDCS — For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional training task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the training task ends.
Device: Sham-tDCS — For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued. Participants will also receive the twenty-minute executive functional training task five minutes subsequent to the stimulation mode.
Behavioral: Cognitive training — Participants will complete an online cognitive training program consisting of 10 consecutive daily weekday training sessions while they receive either the active or sham tDCS stimulation. Each training session will last for 20 minutes. The online cognitive training program will comprise five exercises assessing information processing speed and executive function capacities. Each exercise will take approximately 4 minutes to complete. Given many studies, across different neurological/neuropsychiatric diagnoses, especially for people with autism, it has long been established that social skills and functioning are closely related, and multiple studies have shown that executive function training can improve social functioning in autism or vice versa (i.e. social skills training improves executive functioning in autism), it is reasonable to include cognitive training in this tDCS protocol.

SUMMARY:
Autism spectrum disorder (ASD) is a pervasive and lifelong developmental disorder that currently affects 1 in 54 children. Individuals with autism are often severely impaired in communication, social skills, and cognitive functions. Particularly detrimental characteristics typical of ASD include the inability to relate to people and the display of repetitive stereotyped behaviors and uncontrollable temper outbursts over trivial changes in the environment, which often cause emotional stress for the children, their families, schools and neighborhood communities. To date, there is no cure for ASD, and the disorder remains a highly disabling condition. Recently, transcranial direct current stimulation (tDCS), a noninvasive neuromodulation technique, has shown great promise as an effective and cost-effective tool for reducing core symptoms, such as anxiety, aggression, impulsivity, and poor social communication, in patients with autism. Although the empirical findings in patients with ASD are encouraging, it remains to be determined whether these experimental data can be translated into real-world benefits. An important next step is to better understand the factors affecting the long-term efficacy of tDCS treatment - in particular, the possible risk factors associated with relapse in patients with ASD and the role of booster session tDCS as an add-on treatment to induce long-lasting neuroplastic effects in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are confirmed by a clinical psychologist based on the Diagnostic and Statistical Manual of Mental Disorders-5th Ed (DSM-V) criteria of Autism spectrum disorder and structured interview with their parents or primary caregivers on their developmental history using the Autism Diagnostic Interview-Revised (ADI-R).
* Individuals with ASD who are comorbid with ADHD symptoms will be included if they were willing to abstain from the use of these medications at least 96 hours before the commencement, until the completion, of the treatment.
* In view of the fact that neuroadaptation to antipsychotics typically occurs within six months, potential participants who are prescribed antipsychotic medications will only be included if the dosage of the medication remained unchanged for six months or more before the experimental period.

Exclusion Criteria:

* Individuals without a confirmed diagnosis from the clinical psychologist, with a history of other neurological and psychiatric disorders and head trauma, or on psychiatric medication will be excluded from the study.
* In view of the possibility of seizure induction by tDCS, potential ASD participants comorbid with epilepsy will be excluded.
* Potential participants comorbid with mood or anxiety disorders will also be excluded.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in social responsiveness - Social Responsiveness Scale-2nd edition (SRS-2) | First day of intervention, 1-month, 3-month, 6-month and 12-months after treatment (5 time points)
  SRS-2 is a sensitive measure of social functioning in children that detects even subtle symptoms that are highly related to ASD. It uses a four-point scale and focuses on different aspects of socialization. The total score reflects the clinical effectiveness of tDCS, and higher scores indicate greater symptom severity. It has been shown that SRS-2 is sensitive to detect changes in social communication improvement related to improved cognitive functioning after treatment. SRS-2 assessments will be conducted before and immediately after tDCS treatment.

SECONDARY OUTCOMES:
tDCS safety and clinical response in tDCS outcome | First day of intervention, 1-month, 3-month, 6-month and 12-months after treatment (5 time points)
  To assess tDCS safety, participants will be asked to complete an adverse effects questionnaire (AEQ) which charts the presence of uncomfortable sensations and changes emotions, cognition and perceptions.
  Based on the tDCS outcome recorded immediately after tDCS treatment, participants will be categorized into responders and non-responders based on the percentage of change in the total SRS score. Participants who show reductions of at least 10% in total SRS scores as compared to baseline scores will be considered responders. This percentage reduction benchmark was set with reference to the minimal clinically important difference (MCID) and calculated using the standard error measurement method from an ASD sample in a previous randomized controlled trial.
Change in neuropsychological measures - CANTAB® cognitive tests | First day of intervention, 1-month, 3-month, 6-month and 12-months after treatment (5 time points)
  Cambridge Neuropsychological Test Automated Battery (CANTAB®) includes computerized tests that are correlated to neural networks and have demonstrated high sensitivity in detecting changes in neuropsychological performance. The tests in this battery-the Reaction Time (RTI), Spatial Working Memory (SWM), and Multitasking Tests (MTT)-are well validated and are highly sensitive to the core domains impaired in patients with ASD, including to response/reaction time, working memory, attention, inhibition, and cognitive flexibility.
Change in EEG E/I ratio measurement | First day of intervention, 1-month, 3-month, 6-month and 12-months after treatment (5 time points)
  Each participant will be tested individually using the Starstim 32 hybrid EEG/tCS device (Neuroelectrics®) to collect EEG data. EEG measurements will be taken in the resting state before and immediately after the 10-session intervention program. Participants will be instructed to sit still and focus their attention on a "+" displayed on a computer monitor during eyes-open resting conditions for 5 minutes. Raw data will be processed with the EEGLAB Toolbox using MATLAB® R2019a (The MathWorks Inc., Natick, Massachusetts, USA). Data from 19 electrode positions (Fp1, Fp2, F3, F4, F7, F8, Fz, T3, T4, T5, T6, C3, C4, Cz, P3, P4, Pz, O1, and O2) will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Han, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong